CLINICAL TRIAL: NCT06428292
Title: Comparison of the Effects of Fully Immersive Virtual Reality in Combination With Treadmill and Bicycle on Functional Capacity in Children With Cerebral Palsy
Brief Title: Fully Immersive Virtual Reality Applications in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Ayhan (Other)
Responsible Party: Sponsor-Investigator, Omer Ayhan, Principal investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC-FTR-OA-01
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: Virtual Reality; Function; Balance; Physical Therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator administering the treatment and the investigator performing the evaluations will be different. The evaluator will not know about the interventions that the participants received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined treadmill with virtual reality (Active Comparator): Combining a virtual reality device with a treadmill and using it in a virtual environment, allowing the person to walk in different virtual environments
  Interventions: Device: Virtual reality device branded ''Meta Quest 2''
- stationary bike combined with virtual reality (Active Comparator): Combining a virtual reality device with a stationary bike and using it in a virtual environment, allowing the person to walk in different virtual environments
  Interventions: Device: Virtual reality device branded ''Meta Quest 2''

INTERVENTIONS:
Device: Virtual reality device branded ''Meta Quest 2'' — Combining different exercise equipment with a virtual reality device and using them in a virtual environment can be used to decide which one is more effective.

SUMMARY:
This study was conducted in children diagnosed with Cerebral Palsy (CP); It is a prospective randomized clinical study planned to examine the effects of treadmill and bicycle ergometer applications combined with fully immersive virtual reality (TISG) on motor function, balance and walking.

DETAILED DESCRIPTION:
The aim of this study is in children diagnosed with Cerebral Palsy (CP); It is a comparative study of the effects of treadmill and bicycle ergometer applications combined with total immersive virtual reality (TISG) on motor function, balance and walking. 34 cases diagnosed with Cerebral Palsy between the ages of 12-18 and attending a rehabilitation center will be included in the study. The sample will be divided into two groups by randomization (TİSG combined with treadmill group n = 17, TİSG combined with bicycle ergometer group = 17). Evaluations will be made before and at the end of treatment. An exercise program that will last 45 minutes twice a week for six weeks will be applied to both study groups. The treadmill combined with TİSG group will be given walking training on the treadmill in a virtual environment using virtual reality glasses. The TISG and combined bicycle ergometer group will be given exercise training on the bicycle ergometer in a virtual environment using virtual reality glasses. For both groups, this process will continue in the same order for each exercise in the session. It is assumed that performing the bicycle ergometer in a sitting position makes this exercise safe, easier to perform, and can be performed at different levels of motor function, regardless of the severity of motor impairment. Based on this assumption, this study aimed to compare the use of bicycle ergometer combined with TISG with the treadmill combined with TISG in improving functional capacity, balance and walking functions in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with spastic cerebral palsy
* Being between the ages of 12 - 18
* Being at Level 1 and 2 according to the Gross Motor Function Classification System (GMFSS)
* Being able to understand and speak Turkish
* Not using medical treatment (including botox) in the last six months
* No visual or auditory problems that would hinder communication during applications.
* Having the cognitive skills to adapt to the application and application controls where the intervention is required.

Exclusion Criteria:

* Presence of secondary orthopedic and neurological problems/problems that are severe enough to affect participation in the study (advanced joint instability, severe scoliosis, nystagmus, etc.).
* Having a neurodegenerative disease that may cause attacks during virtual reality applications
* Presence of epilepsy
* Having undergone lower extremity surgery within the last year
* Presence of hypersensitivity to visual stimuli
* Development of vestibular problems with the use of virtual reality devices

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure - 88 | 2 times in 8 weeks
  Gross Motor Function Measure - 88 is a well-known scoring system that evaluates changes in gross motor function. Gross Motor Function Measure - 88 has no age limit and is divided into five gross motor function dimensions: (A) lying and rolling, (B) sitting, (C) crawling and kneeling, (D) standing, and (E) walking, running and jumping. It consists of 88 items. Each item is scored on a 4-point scale (0-1-2-3). A higher score means better motor function.
6 Minute Walk Test | 2 times in 8 weeks
  6 Minute Walk Test is a standardized, inexpensive and easy-to-implement walking test in which the distance walked in 6 minutes is measured under controlled conditions, the person determines his/her own pace. 6 Minute Walk Test is commonly used to assess functional capacity in children with cerebral palsy (CP)

SECONDARY OUTCOMES:
10 Meter Walk Test | 2 times in 8 weeks
  It is a test used to evaluate the walking speed of individuals. They walk at their normal speed, with or without assistance, on a 14-meter walkway, and the time required for each participant to cover a 10-meter walking distance is measured, starting from 2 marked points 2 m after the starting point and 2 m before the end point.
Timed Up And Down Stairs Test | 2 times in 8 weeks
  Timed Up and Down Stair Test attempts to obtain information about the individual's functional mobility by evaluating how long it takes to ascend and descend a 14-step staircase.
Timed Up and Go Test | 2 times in 8 weeks
  Timed Up and Go Test is a valid and reliable test method used to evaluate functional mobility and static and dynamic balance in children with CP. Participants have to stand up from a chair without armrests from the starting position with hips, knees and ankles bent at 90°, walk 3 meters, and return. and they are asked to sit on the chair. Completing the test in less time means more mobility.
Gross Motor Function Classification System | 2 times in 8 weeks
  Gross Motor Function Classification System was developed to measure the 'severity of movement disability' in children with cerebral palsy (CP). Gross Motor Function Classification System provides a method to classify the functional abilities of children with CP into one of five levels. As the grade level approaches five, it means that the child's functional ability decreases and he becomes more dependent.
Pediatric Berg Balance Scale | 2 times in 8 weeks
  The Pediatric Berg Balance Scale, a modified version of the Berg Balance Scale, is a 14-item, criterion-referenced measurement method that examines functional balance in the context of daily tasks. The 14 items that make up the Pediatric Berg Balance Scale are scored on a 4-point scale. A higher score means better balance.

CONTACTS AND LOCATIONS:
Overall Officials: Ipek Yeldan, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul Ünivesitesi - Cerrahpaşa, Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ochandorena-Acha M, Terradas-Monllor M, Nunes Cabrera TF, Torrabias Rodas M, Grau S. Effectiveness of virtual reality on functional mobility during treadmill training in children with cerebral palsy: a single-blind, two-arm parallel group randomised clinical trial (VirtWalkCP Project). BMJ Open. 2022 Nov 3;12(11):e061988. doi: 10.1136/bmjopen-2022-061988. PMID 36328390
- [Background] Cho C, Hwang W, Hwang S, Chung Y. Treadmill Training with Virtual Reality Improves Gait, Balance, and Muscle Strength in Children with Cerebral Palsy. Tohoku J Exp Med. 2016 Mar;238(3):213-8. doi: 10.1620/tjem.238.213. PMID 26947315
- [Background] Zeng N, Pope Z, Gao Z. Acute Effect of Virtual Reality Exercise Bike Games on College Students' Physiological and Psychological Outcomes. Cyberpsychol Behav Soc Netw. 2017 Jul;20(7):453-457. doi: 10.1089/cyber.2017.0042. PMID 28715263
- [Background] Gagliardi C, Turconi AC, Biffi E, Maghini C, Marelli A, Cesareo A, Diella E, Panzeri D. Immersive Virtual Reality to Improve Walking Abilities in Cerebral Palsy: A Pilot Study. Ann Biomed Eng. 2018 Sep;46(9):1376-1384. doi: 10.1007/s10439-018-2039-1. Epub 2018 Apr 27. PMID 29704186